CLINICAL TRIAL: NCT02995343
Title: Evaluation of the Ovarian Reserve in Patients Who Hypogastric Arteries and or Uterine Arteries Had Been Ligated
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Cagdas Sahin, MD, Ege University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2.100.2014.0076
Record Dates: First submitted 2016-12-12; First posted 2016-12-16 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Ovarian Reserve; Hypogastric Artery Ligation; Uterine Artery Ligation

ARMS (2):
- Hypogastric and/or uterine artery ligation (Experimental): Patients who had been ligated hypogastric artery and or uterine artery for ceasing uterine bleeding during c-section
  Interventions: Procedure: Hypogastric and/or uterine artery ligation
- Normal postpartum women (No Intervention)

INTERVENTIONS:
Procedure: Hypogastric and/or uterine artery ligation
  Arms: Hypogastric and/or uterine artery ligation

SUMMARY:
Patients who hypogastric arteries and/or uterine arteries had been ligated will be evaluated in terms of ovarian reserve markers such as anti-mullerian hormone levels, ovarian volumes, antral follicule count, follicule stimuli hormone and estrogen levels. Investigators will search their archives for finding suitable patients for study. Investigators will especially notice being at least 6 month time of interval between surgery and evaluation time. Ultrasound examination and taking blood sample will be performed on 2nd or 3th day of menstrual cycle. These results will be compared with normal postpartum women's results. It will be evaluated that there is or not any effect of the hypogastric arteries and/or uterine arteries on ovarian reserve

ELIGIBILITY:
Inclusion Criteria:

* Patients had been ligated hypogastric and/or uterine arteries
* Patients are in 6 month period after surgery
* Without performed hysterectomy
* No older than 40 years old
* No history about endocrinopathy which have an effect upon ovarian reserve

Exclusion Criteria:

* Patients had been made other gynecologic surgery such as fallopian tube ligation and hysterectomy etc.
* Patients are older than 40 years old
* Patients use drugs which have an effect upon ovarian reserve
* Patients have diseases which have an effect upon ovarian reserve such as some endocrinopathy, malign diseases which require radiotherapy and chemotherapy etc.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Anti-mullerian hormone levels will be evaluated | 6 months after surgery and delivery
Antral Follicule Count will be evaluated | 6 months after surgery and delivery
Ovarian volume will be evaluated | 6 months after surgery and delivery
Follicule Stimuli Hormone levels will be evaluated | 6 months after surgery and delivery
Estrogen levels will be evaluated | 6 months after surgery and delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Medicine Faculty, Department of Obstetrics and Gynecology, Izmir, Turkey (Türkiye)